CLINICAL TRIAL: NCT04083131
Title: Sense of Coherence and Primary Dysmenorrhea in High School Girls in Finistere: Cross-sectional Observational Study
Brief Title: Sense of Coherence and Primary Dysmenorrhea in High School Girls in Finistere, France
Acronym: DysM et SOC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: DysM et SOC (29BRC19.0112)
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Primary Dysmenorrhea
Keywords: Sens of coherence; Primary dysmenorrhea; Salutogenesis; Teenagers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the relation between sens of coherence and primary dysmenorrhea. Aself-questionnaire is completed by a sample of girls aged between 14 and 19, schooled in Finistère (France).

DETAILED DESCRIPTION:
Primary dysmenorrhea affects more than 60% of adolescent girls. Menstrual pain increases absenteeism and lowers self-esteem and academic performance. Moreover, dysmenorrheal women suffer more depression and anxiety.

Sense of coherence (SOC) is composed of three items:

* comprehensibility: what the person understands about his illness
* manageability: what the person does to cope
* meaningfulness: what the disease means to the person. A high SOC score is related to good mental and physical health. The aim of this study will be to determine if there is a relationship between primary dysmenorrhea and the sense of coherence.

A self-questionnaire composed of the SOC-13 and a scale evaluating dysmenorrhea will be proposed in the voluntary high schools of Finistère (France) to the girls of the classes chosen at random.

ELIGIBILITY:
Inclusion Criteria:

* student in high schools
* aged 14 and 19 years
* with menstrual cycle

Exclusion Criteria:

* Illiteracy
* student and parents opposition

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: High school girls in Finistère
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Presence / absence of dysmenorrhea | Inclusion - Day 0
  Presence / absence of dysmenorrhea objectified by Visual Analogue Scale (EVA) from 0 to 10 indicating the average pain over the last 3 cycles (if greater than 3 without treatment = primary dysmenorrhea)
Sense of coherence | Inclusion - Day 0
  Sense of coherence measured by the self-administered French SOC-13 questionnaire (Likert scale).

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Lycée de l'Harteloire, Brest
  - Lycée Jean-Marie Le Bris, Douarnenez
  - Lycée de l'Elorn, Landerneau
  - Lycée du Léon, Landivisiau
  - Lycée Brizeux, Quimper
  - Lycée Roz Glas, Quimperlé

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 6 months and ending three years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.